CLINICAL TRIAL: NCT03578068
Title: Translation and Validation of the French Version of the Postoperative Quality of Recovery Score QoR-15
Acronym: QoR-15F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7051
Record Dates: First submitted 2018-05-28; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-05

CONDITIONS: Recovery of Function
Keywords: Quality of Recovery; Postoperative; Surgery; French; Translation; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After a surgery, the recovery of the previous health status of patients, such as walk, body care, sleep, diet, feeling of comfort, is one of the priorities of the perioperative medicine. The QoR-15 was designed to measure quality of recovery after surgery. It provided a valid, extensive and efficient evaluation of the postoperative quality of recovery. The primary objectives of this study is to translate the original QoR-15 questionnaire into French, and do a full psychometric evaluation of the French version. We will test its validity, reliability, responsiveness, and clinical acceptability and feasibility, with patients undergoing abdominal, orthopedic, […], gynecological surgery, in the University Hospital of Strasbourg. The secondary objectives will be to evaluate the quality of recovery of the patients who undergone surgery at Strasbourg University Hospital, and to evaluate the incidence of postoperative complications occurring within three months postoperatively and a possible association with the QoR-15F.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient operated at Strasbourg University Hospital for a minor, intermediate or major programmed surgery
* Patient agreeing to use his data for research purposes

Exclusion Criteria:

* Patient operated on a surgery for which it is highly probable that the postoperative management does not allow him to propose the completion of the J1 questionnaire
* Patient unable to express non-opposition to participation in the study
* Patient expressing opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient operated at Strasbourg University Hospital for a minor, intermediate or major programmed surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
QoR-15F score Title: QoR-15F score Description: Time Frame: 24h befor surgery Outcome 2 Title: QoR-15F score Description: Time Frame: 24h after surgery | 24h after surgery
  the score is calculated from the questionnaire 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Noll, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service D'Anesthesiologie - Reanimation Chirurgicale, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demumieux F, Ludes PO, Diemunsch P, Bennett-Guerrero E, Lujic M, Lefebvre F, Noll E. Validation of the translated Quality of Recovery-15 questionnaire in a French-speaking population. Br J Anaesth. 2020 Jun;124(6):761-767. doi: 10.1016/j.bja.2020.03.011. Epub 2020 Apr 15. PMID 32303379